CLINICAL TRIAL: NCT04246892
Title: Impact of Alarm Reduction on Delirium in ICU
Acronym: ALADIN
Status: Terminated | Type: Observational
Why Stopped: technical problem, no change of the monitors in the ICU ward
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Lev VOLKOV, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2019PI225
Record Dates: First submitted 2020-01-20; First posted 2020-01-29 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group before alarm withdrawal
- groupe after alarm withdrawal

SUMMARY:
Delirium is an acute and fluctuating disturbance of consciousness and can occur in 80% of critically ill patients. Delirium is more frequent in mecanically ventilated patients and is associated with longer hospital stay, increased cognitive impairment and mortality. On the occasion of the change of the monitors in the ICU ward, allowing a total withdrawal of alarms in patients room, this study evaluates the prevalence of delirium before and after the alarm withdrawal. During the first period the patients will be monitored as usual, and during the second period patients will be monitored without alarms ringing in patients room. Delirium will be screened with a validated, clinical tool.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years, admission to ICU

Exclusion Criteria:

* length of stay in ICU<24 hours, moribund patient, deafness, dementia, psychiatric pathology, delirium at admission, acute neurological pathology at admission (stroke, epilepsy, neuro-infection), hepatic encephalopathy, admission for cardiac arrest, admission for voluntary drug intoxication, pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients admitted to ICU, and who meet inclusion criteria
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
prevalence of delirium, according to a ICDSC score>3 | at the end on the ICU stay, an average of 6 days
  prevalence of delirium in each group

SECONDARY OUTCOMES:
prevalence of sub-syndromic delirium in each group, according to a ICDSC score<4 and absence of delirium | at the end on the ICU stay, an average of 6 days
length of mecanical ventilation (days) | at the end on the ICU stay, an average of 6 days
length of stay in ICU (days) | at the end on the ICU stay, an average of 6 days
in patients presenting a delirium, duration of delirium (days) defined by the number of days with a ICDSC score>3 | at the end on the ICU stay, an average of 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Lev VOLKOV, Study Director — Central Hospital, Nancy, France
Locations (1):
- CHRU Nancy, Nancy, France